CLINICAL TRIAL: NCT02714660
Title: The Work of Being a Patient: A Mixed Methods Characterization of the Work of Being a Patient With Type 2 Diabetes Mellitus Using Real-time Data Collection Via a Smartphone Application
Brief Title: The Work of Being a Patient With Diabetes: Data Collection Via a Smartphone Application
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Victor Montori, MD, Mayo Clinic
Other Study IDs: 15-005767
Record Dates: First submitted 2016-03-17; First posted 2016-03-21 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Type 2 Diabetes: Adults with type 2 diabetes will be enrolled in this mixed methods observational study.
  Interventions: Other: none, observational study

INTERVENTIONS:
Other: none, observational study

SUMMARY:
This mixed methods study aims to answer the question: "What is the work of being a patient with type 2 diabetes mellitus?" .

DETAILED DESCRIPTION:
This study will describe how much time persons with type 2 diabetes mellitus spend on health management and the burden they experience from these activities.

ELIGIBILITY:
Inclusion Criteria:

* receiving medical care at Mayo Clinic endocrine subspecialty clinic
* diagnosis of type 2 diabetes

Exclusion Criteria:

* unable to provide consent
* patients who reside in an extended care of intermediate care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type 2 diabetes with receiving care at Mayo Clinic endocrinology department.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Mean Score on Burden of Treatment Questionnaire | Baseline
  The 48-item version of the Patient Experience with Treatment and Self-Care (PETS)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Montori, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No